CLINICAL TRIAL: NCT06217484
Title: Investigation of Effects of Delayed Feedback on Non-motor Symptoms in Individuals With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Ekaterina Dobryakova, Assistant Director of Neuroscience Research, Kessler Foundation
Other Study IDs: E-1228-23
Record Dates: First submitted 2023-12-28; First posted 2024-01-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; learning; feedback
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parkinson Disease: Participants with Parkinson Disease; Single group.
  Interventions: Behavioral: delayed feedback

INTERVENTIONS:
Behavioral: delayed feedback — participants learn through either immediate or delayed feedback during a computer task

SUMMARY:
Learning deficits are frequent in individuals with Parkinson's Disease. Clear feedback is integral because through feedback individuals know whether they should stick with an action that they have been doing (if the feedback is positive), or change their course of action (if the feedback is negative). Learning though immediate feedback has been shown to be depended on the brain chemical dopamine that is disrupted in individuals with Parkinson's Disease. During learning, feedback can also be presented after a delay. The investigators propose that learning through delayed feedback will lead to greater learning in individuals with Parkinson's Disease, since learning through delayed feedback does not rely on dopamine. During the proposed paradigm, participants with Parkinson's Disease complete a multiple-choice test. After making their selection on the multiple-choice test, they either see feedback immediately or are given feedback 25 minute later after reviewing their selection on the multiple-choice test. The investigators hypothesize that participants will learn better when they are provided with delayed feedback.

ELIGIBILITY:
Inclusion Criteria:

* Only participants with scores above 24/30 on the Montreal Cognitive Assessment will be recruited for participation to exclude dementia.

Exclusion Criteria:

* Individuals with neurological conditions other than PD such as epilepsy, multiple sclerosis, brain tumors, etc. will be excluded to control for the effects these conditions have on the brain and behavior.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Parkinson Disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Percent correct responses will be collected through the computer software | testing lasts 60 minutes and completed in 1 day
  Response accuracy per trial

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Dobryakova, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No